CLINICAL TRIAL: NCT02375802
Title: A Pilot Study: Evaluating the Safety and Feasibility of Using Autologous Adipose-Derived Stromal Cells From Stromal Vascular Fraction (SVF) on Adults With Pressure Ulcers or Diabetic Foot Ulcers
Brief Title: Adipose-Derived Stromal Cells (ASC's) for Pressure Ulcers
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Houssam Farres, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-002855
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pressure Ulcer
Keywords: Stem cells
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Liposuction will be done to extract 50-100 cc of adipose tissue which will be processed to obtain the stromal cells. The adipose-derived stromal cells will be injected into a fibrin sealant applicator and applied to the wound (intervention), Patients will receive 5.0x106 ASCs per cubic centimeter of wound area. The wound will be dressed with an occlusive dressing and soft silicone dressing. The dressing will remain in place for one week (minimally, 3 days). Follow-up will occur weekly for 6 weeks.
  Interventions: Biological: Adipose-derived stromal cells; Drug: Adipose-derived stromal cells

INTERVENTIONS:
Biological: Adipose-derived stromal cells — Adipose-derived stromal cells contain stem cells which have been successful in enhancing wound healing. The product used as the carrier is a fibrin sealant called TISSEEL. Pre-pilot testing was done to verify viability of the stromal cells for up to 72 hours in the fibrin sealant.
  Other Names: ASC's
Drug: Adipose-derived stromal cells

SUMMARY:
This pilot study of 12 patients will test the safety and efficacy of applying autologous, adipose-derived stromal cells (ASCs), uncultured, on a Stage III or IV pressure ulcer or diabetic foot ulcers. Patients will undergo a minimal risk liposuction procedure to withdraw 50-100 cc of adipose tissue. The tissue would be processed to extract the stromal layer of cells that contain stem cells. The ASCs would be injected into a fibrin sealant to be applied to the wound. Patients would be followed for 6 weeks to assess wound healing and tolerance of the treatment.

DETAILED DESCRIPTION:
Wound healing for Stage III and IV pressure ulcers or diabetic foot ulcers can take four to six weeks or longer and cost upwards of $40,000 to treat. Past studies have shown that adipose tissue contains progenitor cells or regenerative cells that can release multiple angiogenic growth factors and cytokines including vascular endothelial growth factor (VEGF), hepatocyte growth factor (HGF) and chemokine stromal cell-derived factor-1 (SDF-1). A current literature review revealed that there is research related to use of stem cells to enhance wound healing, in particular with ischemic or radiation-induced ulcers. However, there is limited research completed on use of stem cells or ASCs with pressure ulcers. The goal is to heal pressure ulcers faster and prevent further complications using the patient's own natural ASCs.

ELIGIBILITY:
Inclusion Criteria

* Males and females
* Stage III pressure ulcers measuring 5 cc - 36 cc in volume (as measured by filling the wound with Normal Saline).
* Inpatient or outpatient treatment of pressure ulcers
* Diabetic Foot Ulcer Stage 1 or 2 of any size
* Co-morbidities may include:

  * Peripheral Vascular Disease (PVD)
  * Coronary Artery Disease (CAD)
  * Chronic Renal Disease (CRD)
  * Chronic Liver Disease (CLD)
  * Hypertension (HTN)
  * Diabetes
* The ability of subjects to give appropriate consent or have an appropriate representative available to do so
* The ability of subjects to return for weekly wound assessments

Exclusion Criteria

* Patients with allergies to TISSEEL, Tegaderm, or silicon
* Diabetics with poor glucose metabolic control (HbA1c > 9)
* Target wounds that are in close proximity to potential cancerous lesions
* Patients who require Negative Pressure Wound Therapy (NPWT), limb amputation, or surgical intervention at the target wound at the time of screening
* Wounds located on the face
* Patients with Stage 5 or 6 Peripheral Vascular disease (specifically, wounds that are caused by peripheral vascular disease such as leg ulcers)
* Wounds caused by diabetes mellitus (diabetic foot ulcers).
* BMI of <16 Clinical signs of critical colonization or local infection
* Prolonged (> 6 months) use of steroids
* Patients on active regimen of chemotherapy
* Patients receiving radiation in proximity of wound
* Decompensated chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-07; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Free of wound infection | one week
  Symptoms include fever along with new or increasing pain, erythema, local warmth, swelling, purulent discharge, and/or malodor

SECONDARY OUTCOMES:
Liposuction procedure without complication | one week
  Signs of adverse reactions to the liposuction procedure include an allergy to the Hunstad solution, infection at the puncture wound site or risk of bleeding at the puncture wound site. Risks include bleeding or infection at the site and bruising for approximately one week. No adverse consequences of fluid overload have been associated with low volume liposuction.
Improved wound healing | weekly observation for 6 weeks
  Wound healing is greater than 20% healing within two weeks documented by measurement of the wound bed or wound healing to less than the dermal layer documented by photography and agreement of healing between research nurse and wound physician consultant. Would not expect deterioration to a more severe level of tissue injury

CONTACTS AND LOCATIONS:
Overall Officials: Houssam Farres, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu D, Chen B, Liang Z, Deng W, Jiang Y, Li S, Xu J, Wu Q, Zhang Z, Xie B, Chen S. Comparison of bone marrow mesenchymal stem cells with bone marrow-derived mononuclear cells for treatment of diabetic critical limb ischemia and foot ulcer: a double-blind, randomized, controlled trial. Diabetes Res Clin Pract. 2011 Apr;92(1):26-36. doi: 10.1016/j.diabres.2010.12.010. Epub 2011 Jan 8. PMID 21216483
- [Background] Bura A, Planat-Benard V, Bourin P, Silvestre JS, Gross F, Grolleau JL, Saint-Lebese B, Peyrafitte JA, Fleury S, Gadelorge M, Taurand M, Dupuis-Coronas S, Leobon B, Casteilla L. Phase I trial: the use of autologous cultured adipose-derived stroma/stem cells to treat patients with non-revascularizable critical limb ischemia. Cytotherapy. 2014 Feb;16(2):245-57. doi: 10.1016/j.jcyt.2013.11.011. PMID 24438903
- [Background] Rigotti G, Marchi A, Galie M, Baroni G, Benati D, Krampera M, Pasini A, Sbarbati A. Clinical treatment of radiotherapy tissue damage by lipoaspirate transplant: a healing process mediated by adipose-derived adult stem cells. Plast Reconstr Surg. 2007 Apr 15;119(5):1409-1422. doi: 10.1097/01.prs.0000256047.47909.71. PMID 17415234
- [Result] Akita S, Yoshimoto H, Akino K, Ohtsuru A, Hayashida K, Hirano A, Suzuki K, Yamashita S. Early experiences with stem cells in treating chronic wounds. Clin Plast Surg. 2012 Jul;39(3):281-92. doi: 10.1016/j.cps.2012.04.005. Epub 2012 May 22. PMID 22732376
- [Result] Bourin P, Bunnell BA, Casteilla L, Dominici M, Katz AJ, March KL, Redl H, Rubin JP, Yoshimura K, Gimble JM. Stromal cells from the adipose tissue-derived stromal vascular fraction and culture expanded adipose tissue-derived stromal/stem cells: a joint statement of the International Federation for Adipose Therapeutics and Science (IFATS) and the International Society for Cellular Therapy (ISCT). Cytotherapy. 2013 Jun;15(6):641-8. doi: 10.1016/j.jcyt.2013.02.006. Epub 2013 Apr 6. PMID 23570660
- [Result] Falanga V, Iwamoto S, Chartier M, Yufit T, Butmarc J, Kouttab N, Shrayer D, Carson P. Autologous bone marrow-derived cultured mesenchymal stem cells delivered in a fibrin spray accelerate healing in murine and human cutaneous wounds. Tissue Eng. 2007 Jun;13(6):1299-312. doi: 10.1089/ten.2006.0278. PMID 17518741
- [Result] Gorecki C, Brown JM, Nelson EA, Briggs M, Schoonhoven L, Dealey C, Defloor T, Nixon J; European Quality of Life Pressure Ulcer Project group. Impact of pressure ulcers on quality of life in older patients: a systematic review. J Am Geriatr Soc. 2009 Jul;57(7):1175-83. doi: 10.1111/j.1532-5415.2009.02307.x. Epub 2009 May 21. PMID 19486198
- [Result] Graves N, Birrell F, Whitby M. Effect of pressure ulcers on length of hospital stay. Infect Control Hosp Epidemiol. 2005 Mar;26(3):293-7. doi: 10.1086/502542. PMID 15796283
- [Result] Kim I, Lee SK, Yoon JI, Kim DE, Kim M, Ha H. Fibrin glue improves the therapeutic effect of MSCs by sustaining survival and paracrine function. Tissue Eng Part A. 2013 Nov;19(21-22):2373-81. doi: 10.1089/ten.TEA.2012.0665. Epub 2013 Jul 16. PMID 23701237
- [Result] Sarasua JG, Lopez SP, Viejo MA, Basterrechea MP, Rodriguez AF, Gutierrez AF, Gala JG, Menendez YM, Augusto DE, Arias AP, Hernandez JO. Treatment of pressure ulcers with autologous bone marrow nuclear cells in patients with spinal cord injury. J Spinal Cord Med. 2011;34(3):301-7. doi: 10.1179/2045772311Y.0000000010. PMID 21756569
- [Result] Teraa M, Sprengers RW, van der Graaf Y, Peters CE, Moll FL, Verhaar MC. Autologous bone marrow-derived cell therapy in patients with critical limb ischemia: a meta-analysis of randomized controlled clinical trials. Ann Surg. 2013 Dec;258(6):922-9. doi: 10.1097/SLA.0b013e3182854cf1. PMID 23426345
- [Result] Zimmerlin L, Rubin JP, Pfeifer ME, Moore LR, Donnenberg VS, Donnenberg AD. Human adipose stromal vascular cell delivery in a fibrin spray. Cytotherapy. 2013 Jan;15(1):102-8. doi: 10.1016/j.jcyt.2012.10.009. PMID 23260090
- [Result] Cherubino M, Rubin JP, Miljkovic N, Kelmendi-Doko A, Marra KG. Adipose-derived stem cells for wound healing applications. Ann Plast Surg. 2011 Feb;66(2):210-5. doi: 10.1097/SAP.0b013e3181e6d06c. PMID 21200308